CLINICAL TRIAL: NCT07224269
Title: A Pilot Study of the Effect of Terazosin on ATP Levels in People With Amyotrophic Lateral Sclerosis
Brief Title: Effect of Terazosin on ATP Levels in People With Amyotrophic Lateral Sclerosis
Acronym: TZ-ALS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Andrea Swenson, Clinical Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202408197
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis; Adenosine Triphosphate Activities
Keywords: amyotrophic lateral sclerosis; open label; terazosin; clinical trial
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Terazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Terazosin (Experimental)
  Interventions: Drug: Terazosine

INTERVENTIONS:
Drug: Terazosine — Titrating up to 5 mg PO at bedtime. Trial participants will take terazosin for 12 weeks.

SUMMARY:
This will be a single center, open label pilot study to assess the safety and tolerability of terazosin (TZ) at a dose of 5 milligrams (mg) per os (PO) daily for patients with amyotrophic lateral sclerosis (ALS). The primary outcome of this study is to determine whether TZ increases adenosine triphosphate (ATP) levels in ALS. The investigators will measure adverse outcomes, safety, and tolerability of taking TZ. Procedures include blood draws, spirometry, lumbar punctures, fluorodeoxyglucose-positron emission tomography (FDG-PET) scans, questionnaires, and physical examinations. TZ will be titrated up to 5 mg PO daily. This is a pilot study and is not powered to assess efficacy of this medication. The investigators' hope is that this study will guide future studies of this (and similar) medications for the disease modification of ALS. This study also aims to learn more about how patients produce and use energy and if TZ can help to reverse energy deficits that appear in ALS.

ELIGIBILITY:
INCLUSION CRITERIA

* Ages 18 - 80 years old
* Diagnosed with ALS based on Gold Coast Criteria
* ALS symptom onset within 36 months at enrollment
* Slow vital capacity (SVC) > 65%
* Riluzole use-Never taken or taking a stable dose for at least 4 weeks prior to screening visit or will refrain from starting for the duration of the study
* Edaravone use-Never taken or completed at least one cycle (typically 14 days) prior to screening visit or will refrain from starting for the duration of the study
* Must have the ability to swallow pills at the time of the screening visit, and in the principle investigator's opinion, have the ability to swallow pills for the duration of the study
* Willing to use highly effective contraception for the duration of the trial treatment and for a duration of 80 days after the last dose.

EXCLUSION CRITERIA

* Orthostatic hypotension at screening is defined as decrease in BP > 20 mmHg systolic or > 10 mmHg diastolic and HR increase <20 bpm on transition from supine to sitting or from sitting to standing
* Known allergy or previous adverse reaction to terazosin or related compound
* Current use of terazosin or concurrent use of doxazosin, alfuzosin, prazosin, or tamsulosin at the time of screening visit or within the 3 months prior to baseline visit
* Current diagnosis or healthcare professional-recommended treatment (medication, exercise or diet) of diabetes mellitus (type 1 or type 2)
* Screening glucose >140 mg/dl
* Pregnancy or breastfeeding women
* Taking therapeutic anticoagulant medication (i.e. warfarin, DOAC's, full dose Lovenox or heparin)
* Liver function blood tests (ALT or AST) more than twice the upper limit of normal
* Hemoglobin < 11.0 g/dL
* Traumatic brain injury or post-traumatic stress disorder
* Presence of a confounding acute or unstable medical, psychiatric, or orthopedic condition
* Noncompliant or sporadic use of medications that modulate the central nervous system
* Uncontrolled major depression or bipolar affective disorder, or other mental health disorders that are, in the opinion of the PI, sufficiently severe to increase risk of experiencing an Adverse Drug Reaction (ADR)
* Current suicidal ideation as measured by question 2 of the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Participants with insufficient decisional capacity to provide written informed consent determined by the primary investigator.
* Noncompliant or sporadic use of antihypertensive medications
* Unable to lie supine and still for 60 minutes for the duration of the study
* Contraindications to undergoing lumbar puncture
* Currently taking part in another clinical trial with an investigational medicinal product or having taken part in one in the three months prior to screening visit
* Current diagnosis of diabetes (type 1 or type 2) or healthcare professional-recommended treatment (medication, exercise or diet) of diabetes mellitus
* Screening visit glucose >140 mg/dl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in ATP levels | Baseline and 12 weeks
  Mean percent change from baseline to 12 weeks in whole-blood ATP and brain glycolytic rate using FDG-PET imaging

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Swenson, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No